CLINICAL TRIAL: NCT01907932
Title: Estimation of Spleen Size by Medical Residents With Hand Carried Ultrasound
Brief Title: Estimation of Spleen by Residents With VScan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Graydon Meneilly, Professor, UBC Department of Medicine, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H13-01727
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Splenomegaly
Keywords: splenomegaly; ultrasound; VScan
MeSH Terms: conditions — Splenomegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- normal and various degrees splenomegaly (Experimental): VScan Ultrasound (GE Healthcare, USA) all subjects will be measured by 5 different medical residents
  Each resident will complete questionaire:
  1. Adequacy of image quality
  2. What is best view obtained
  3. Greatest Longitudinal Measure
  4. Diagnosis
  5. Diagnostic Certainty
  6. Time to Complete exam
  Interventions: Device: VScan Ultrasound (GE Healthcare, USA)

INTERVENTIONS:
Device: VScan Ultrasound (GE Healthcare, USA) — VScan Ultrasound used to determine spleen size and the other qualities described in the arm description.
  Other Names: handheld ultrasound (HCU)

SUMMARY:
In internal medicine, assessment of spleen size on physical examination is an extremely important part of the overall evaluation of patients with many illnesses. Examination of the spleen is also one of the core competencies that the investigators expect the students and residents to learn as part of their training. Unfortunately, the sensitivity and specificity of examination of the spleen at the bedside is not very good. The investigators wish to determine if medical residents can be taught to use hand carried ultrasound to accurately assess spleen size. Doing so would make physical examination of the spleen obsolete and transform training objectives for medical trainees.

DETAILED DESCRIPTION:
The diagnosis of splenomegaly is extremely important in managing patients with blood disorders and other medical conditions, such as cirrhosis. The ability to recognize an enlarged spleen in a timely manner can impact patient outcomes. Although the physical exam can be confidently used to diagnosis massive enlargement of the spleen, evaluating lesser degrees of splenomegaly at the bedside proves more difficult. In current practice, the gold standard for diagnosis of splenomegaly is the conventional abdominal ultrasound. The prevalence of splenomegaly in patients with blood conditions and other medical disorders is relatively high. Therefore, the demand for abdominal ultrasound is growing and similarly the cost of caring for patients with these conditions.

In addition, examination of the spleen is one of the core competencies that the investigators expect the students and residents to learn as part of their training. This physical diagnosis maneuver is frequently used to examine residents at the Royal College level and determine their fitness to practice. Unfortunately, the sensitivity and specificity of examination of the spleen at the bedside is not very good.

With the introduction of hand carried ultrasound (HCU) devices, rapid bedside assessment of a patient is now possible. The Visual scan (VScan) (GE Healthcare, USA) allows for 2D imaging on a 3.5 inch display and has shown to have comparable image quality to standard ultrasound for some applications. The VScan and other HCU have been used at point of care to evaluate a number of conditions and can greatly impact treatment decisions in medical patients at the bedside. The ability to recognize splenomegaly in a timely manner can impact patient outcomes. In addition, the use of this technology could significantly impact training standards for students and residents.

It remains unclear whether bedside evaluation with the VScan is able to accurately measure spleen size. The investigators conducted an extensive literature review and the investigators were unable to find any studies attempting to accurately assess spleen size with HCU. The investigators recently demonstrated that trained ultrasonographers can reliably assess spleen size at the bedside using a VScan. The current study aims to determine the diagnostic accuracy of the VScan when used by medical residents who have been trained in its use, in patients with varying degrees of splenomegaly, including normal spleen size. If the investigators can show that medical residents can accurately characterize spleen size at the bedside with a hand carried device, the next stage of the study will be to determine how the investigators can integrate HCU with physical examination at the bedside to assess spleen size.

Design, Specification of Endpoints, and Procedures:

The investigators propose a validation study in 50 patients who have medical conditions that may result in varying degrees of splenomegaly (including normal spleen size) and who are looked after in the hematology clinics at Vancouver General Hospital (VGH). Patients will be recruited based on information provided in the charts in the private offices of hematologists at VGH.

The investigators will also enroll 20 first year medical residents. First year residents will be sent a letter by email describing the study.

Each medical resident will undergo a one hour training sessions by an ultrasonographer regarding the use of HCU to assess spleen size. At the end of the session, they will be evaluated by the sonographer to make sure they know how to use the HCU to acquire images of the spleen. If they are not proficient they will undergo a subsequent one hour training session. On a separate day, a trained ultrasonographer will perform a conventional ultrasound on each patient to accurately measure their spleen size. This information will be provided to the patients hematologist. Subsequently residents will attempt to measure the size of the patient's spleen using the VScan. Each patient will be scanned 5 times by 5 different residents. Each resident will be blinded as to the patient's underlying medical conditions and the results of previous scans. Variables of interest include: adequacy of the study, findings on 2D imaging, overall diagnosis of presence of splenomegaly, confidence level in diagnosis and time to complete test.

The goal is to determine if medical residents can use a hand carried ultrasound device to accurately assess spleen size.

ELIGIBILITY:
Inclusion Criteria:

* patients in the practices of hematologists at VGH who are expected to have normal size spleens as well as various degrees of splenomegaly

Exclusion Criteria:

* will exclude patients who cannot speak English or who cannot give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
longitudinal measure of spleen in centimeters | 1 day

SECONDARY OUTCOMES:
Diagnosis of spleen size | 1 day
  Diagnosis
  1. No Splenic Enlargement
  2. Moderate Splenic Enlargement
  3. Massive Splenic enlargement

OTHER OUTCOMES:
time to complete VScan examination | 1 day
  Time to complete VScan exam
  1. <5min
  2. 5-10 min
  3. 10-15min
  4. >15min
Image quality and best views | 1 day
  Adequacy of study
  1. Image quality inadequate to make diagnosis
  2. Image quality adequate
  3. Image quality excellent Best Views obtained
  a. Supine b. Right Lateral Decubitus
Diagnostic Certainty | 1 day
  Diagnostic Certainty
  1. Not confident
  2. Somewhat confident
  3. Very confident

CONTACTS AND LOCATIONS:
Overall Officials: Graydon S Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health (VCHRI/VCHA), Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No